CLINICAL TRIAL: NCT06636669
Title: The Role of Peri-operative Adjunctive Probiotics in the Prevention of Recurrent Prosthetic Joint Infection of the Hip and Knee
Brief Title: Probiotics in the Prevention of Recurrent Prosthetic Joint Infection of the Hip and Knee
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: American Association of Hip and Knee Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-44452
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Prosthetic-joint Infection; Dysbiosis
Keywords: Probiotics; Hip total joint arthroplasty (TJA); Knee TJA; Recurrent reinfection; DAIR; Surgical site infection (SSI); Patient Reported Outcome Measures (PROMs)
MeSH Terms: conditions — Dysbiosis; Reinfection; Surgical Wound Infection | interventions — Probiotics; Standard of Care

STUDY DESIGN:
Intervention Model Description: A multi-centered, randomized controlled trial (RCT) with two arms will be conducted at two academic, tertiary care centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment- Probiotics and standard of care (Experimental): Participants randomized into this are will receive Culturelle probiotic and standard of care.
  Interventions: Drug: Probiotic; Other: Standard of care
- Controls- Standard of care (Active Comparator): Participants randomized into this are will receive standard of care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Probiotic — Culturelle probiotic, one capsule daily to start following SOC surgical treatment for PJI during the initial 6 weeks of SOC antibiotic treatment.
  Other Names: Culturelle
  Arms: Treatment- Probiotics and standard of care
Other: Standard of care — Standard of care (SOC) treatment includes surgery and antimicrobials.

SUMMARY:
Prosthetic joint infection (PJI) is one of the most devastating complications following total joint arthroplasty (TJA) of the hip and knee. Standard of care (SOC) treatment includes surgery and antimicrobials. Morbidity and mortality remain high despite contemporary treatments. The human body is colonized by billions of organisms, collectively, the microbiome, which is central to healthy immune function. Microbiome disruption, dysbiosis, can impair the immune response to infection.

Despite recent evidence that suggests dysbiosis may be implicated in PJI, the role of probiotics in the treatment of PJI is unknown. Perioperative probiotics have been demonstrated to be safe and effective for infection prevention in abdominal surgery. The investigators hypothesize that perioperative probiotics will reduce re-infection in patients treated for PJI. A multi-centered, randomized controlled trial (RCT) at two academic, tertiary care centers will be conducted to determine the impact of probiotics on recurrent infection following treatment for PJI. Controls will receive SOC; study patients will receive a probiotic, started shortly after the initiation of and for the duration of their antibiotic therapy + 7 days, in addition to SOC. Primary outcome is re-operation for recurrent infection within 1 year.

DETAILED DESCRIPTION:
The primary and secondary aims for this RCT are:

Primary Aim 1.1 To determine the impact of administration of probiotics administered for 6 weeks after the index surgical treatment for PJI on reinfection rates (deep infection) within 1 year following revision TJA for PJI in each of the treatment arms (probiotics and standard of care).

Secondary Aims 2.1 To evaluate the incidence of superficial infections including wound drainage, cellulitis, or infections superficial to the deep fascia within 1 year following revision TJA for PJI in each of the treatment arms (probiotics and standard of care).

2.2 To evaluate the safety of use of probiotics in this population and to monitor the incidence of adverse events in patients administered probiotics versus standard of care in patients undergoing treatment for PJI.

2.3 To evaluate the 1-year mortality rate in patients undergoing revision TJA for PJI in each of treatment arms (probiotics and standard of care).

2.4 To evaluate the rate of wound healing and dehiscence in patients undergoing revision TJA for PJI in each of treatment arms (probiotics and standard of care).

2.5 To evaluate the need for chronic antibiotic suppression for the treatment of PJI at final follow-up of one year following revision TJA for PJI in each of the treatment arms (probiotics and standard of care).

2.6 To evaluate the rate of infection with Clostridium difficile within 90 days of finishing antibiotic therapy in each of the treatment arms (probiotics and standard of care). The risk of developing C. difficile infection is present for 90 days following cessation of antibiotic treatment.

ELIGIBILITY:
All patients scheduled to undergo revision total knee arthroplasty (TKA) or total hip arthroplasty (THA) for infection at the participating institutions will be screened for eligibility in this prospective trial.

Inclusion Criteria:

* Diagnosis of PJI based upon Musculoskeletal Infection Society (MSIS) criteria
* Planned treatment with surgical debridement, antibiotics, implant retention (DAIR), single- and two-stage revision TJA for PJI with an anticipated plan for eventual discontinuation of oral/IV antibiotics.
* Patients with prior PJI in the same joint that has recurred.
* Patients who understand the benefits and risks associated with taking a probiotic and are willing and able to provide informed consent.

Exclusion Criteria:

* Fungal PJI.
* Inflammatory bowel disease, diverticulitis, history of intestinal surgery, or gastrointestinal
* issue where there is concern for gut integrity.
* History of pancreatitis at any point in time.
* History of intolerance to probiotics.
* Immunocompromised patients.
* Revision TJA for aseptic reasons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recurrent Prosthetic Joint Infection (PJI) | 1 year, 2 years after PJI surgery
  The number of participants who develop PJI after PJI surgery will be abstracted from electronic medical records.
Surgical Site Infection (SSI) | 3 months, 6 months, 12 months post PJI surgery
  The number of participants who develop SSI within 12 months of PJI surgery will be abstracted from electronic medical records.

SECONDARY OUTCOMES:
Medical complications | 3 months, 6 months, 12 months post PJI surgery
  This outcome will be assessed from information in the electronic medical records and reported as Yes or No.
Surgical complications | 3 months, 6 months, 12 months post PJI surgery
  This outcome will be assessed from information in the electronic medical records and reported as Yes or No.
Sepsis | 3 months, 6 months, 12 months post PJI surgery
  The number of participants who have a diagnosis of sepsis related to PJI surgery will be abstracted from electronic medical records.
Re-operation for recurrent infection | 3 months, 6 months, 12 months post PJI surgery
  The number of participants who have a re-operation for recurrent infection within 12 months of the PJI surgery will be abstracted from the electronic medical records.
Revision surgery | 3 months, 6 months, 12 months post PJI surgery
  The number of participants who have revision surgery within 12 months of PJI surgery will be abstracted from electronic medical records.
Complications related to the use of probiotics | 3 months, 6 months, 12 months post PJI surgery
  This outcome will be assessed from information in the electronic medical records and reported as Yes or No.
Mortality | 12 months post PJI surgery
  The number of participants who die within 12 months of the PJI surgery will be abstracted from the electronic medical records.
Patient reported health outcomes | 3 months, 6 months, 12 months post PJI surgery
  The Patient-Reported Outcomes Measurement Information System (PROMIS)-10 score ranges from 0 to 20 points, with 0 representing the most severe impairment and 20 representing the best possible health. Low scores may indicate poorer self-reported health and a greater risk of future healthcare utilization.
Patient reported hip disability | 3 months, 6 months, 12 months post PJI surgery
  The Hip disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS, JR) will be used to assess hip disability. It is patient reported and contains 6 items from the original HOOS survey. Items are coded from 0 to 4, none to extreme respectively. HOOS, JR is scored by summing the raw response (range 0-24) and then converting it to an interval score using a table where the interval score ranges from 0 to 100 where 0 represents total hip disability and 100 represents perfect hip health.
Patient reported knee disability | 3 months, 6 months, 12 months post PJI surgery
  Knee Injury and Osteoarthritis Outcome Score, Joint Replacement (KOOS, JR) will be used to assess knee disability. It is patient reported and contains 7 items from the original KOOS survey. Items are coded from 0 to 4, none to extreme respectively. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score using a table.. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Abdeen, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Medical Center, Orthopedic Surgery, Boston, Massachusetts
  - New York University Langone Orthopedics, New York, New York

IPD SHARING:
Plan to Share IPD: No